CLINICAL TRIAL: NCT04491019
Title: Comparison of the Effects of Two Different Exercise Programs on Balance, Posture and Lower Extremity Functions in Obese Adolescents
Brief Title: Comparison of the Effects of Two Different Exercise Programs in Obese Adolescents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Saime Nilay Arman, Assist.Prof., Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 02/10/2019-149844
Record Dates: First submitted 2020-07-27; First posted 2020-07-29 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Obesity, Adolescent
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Balance exercise group (Experimental): Balance exercises will be carried out with a physiotherapist.
  Interventions: Other: Balance exercise group
- Strengthening exercise group (Experimental): Strengthening exercises will be performed with a physiotherapist.
  Interventions: Other: Balance exercise group

INTERVENTIONS:
Other: Balance exercise group — Balance exercises will be carried out with a physiotherapist

SUMMARY:
Obesity is one of the most important health problems of developed and developing countries. Especially in children and adolescents, the prevalence of obesity is increasing at an alarming rate. In obese individuals, the effects of postural control and balance have been reported to cause musculoskeletal problems, and motor control skills have been found to decrease. The aim of this study is to compare the effects of balance exercises and strengthening exercises on balance, posture and lower extremity functions in obese adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 12-18 Body Mass Index to be 95 and above according to percentile values No exercise program in the past 6 months

Exclusion Criteria:

* Having a medical condition that prevents exercise Having a disease of neuromuscular origin Presence of psychiatric or neurological diseases affecting cooperative and cognitive functions Equilibrium effect due to another disease

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-02-27 (Actual); Primary Completion 2020-07-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
The six-minute walking test | Change from baseline to 8 weeks, follow up at two months
  The six-minute walking test is an example of timed distance testing, widely used in clinical research and rehabilitation studies. According to the guidelines published by the American Thoracic Society, 6MWT is an easy-to-use, better tolerated test that reflects daily activities better than other walking tests. It can be applied in a short time. Requires little equipment. The six-minute walk test, used as a field test, is a simple and inexpensive test compatible with daily activities, which does not require exercise equipment. Before starting the test, the patient should rest for at least 10 minutes by sitting in the chair near the starting point. The walking area must be at least 30 m long. A shorter corridor causes more time to be spent for more frequent turns and changes of direction. With the help of stopwatch, it is kept for 6 minutes and the number of laps during the period is calculated and recorded. The functional capacity of the cases will be evaluated with 6MWT.

SECONDARY OUTCOMES:
Sit Up Stand Test | Change from baseline to 8 weeks, follow up at two months
  It reflects the individuals' lower limb muscle strength and functional capacities. For the test, the individual is allowed to sit on the 43.18 cm high chair in the middle of the chair with his back straight, with his feet on the ground and his arms crossed in front of his chest (right hand left shoulder, left hand right shoulder). When the individual is in this position, the test is started with the start command and the number of complete departures that he has made for 30 seconds constitutes the score of the individual. The lower extremity functions of the cases will be evaluated by sit and test.
Evaluation of Muscle Force | Change from baseline to 8 weeks, follow up at two months
  Muscle strength tests are performed to determine the ability to provide strength and stability. One of the methods used in the evaluation of muscle strength is the dynamometer. Compared to isokinetic devices, hand-held dynamometers are considered as a reliable and valid tool for evaluating muscle strength in the clinic due to their easy transportation, cost and small size. The lower extremity muscle strength of the cases will be evaluated with MicroFet 2 brand dynamometer.
10 Step Down Time Test | Change from baseline to 8 weeks, follow up at two months
  All cases are asked to go up to 10 digits (14x28x120 cm) as fast as possible. Step-up time is measured in seconds with a stopwatch. The measurement is repeated three times and the score is recorded by taking the average of the three measurements.
Functional Forward Reach Test | Change from baseline to 8 weeks, follow up at two months
  Functional reach test will be used to evaluate the balance of the cases. The person is asked to stand sideways in a position where the right arm does not touch a tape measure attached to the wall at shoulder height. When the arm is at 90 ° flexion, it is requested to hold the arm in parallel with the tape measure without extending it forward. The distance between the shoulder and the 3rd fingertip is measured. Then, the maximum distance at which he can extend his arm horizontally is measured. The difference between the two positions is calculated in centimeters.
Flamingo Balance Test | Change from baseline to 8 weeks, follow up at two months
  Flamingo Balance Test is used to determine the static balance of the cases. According to this test, the patients stand in balance by standing with the side of the tested side on a wooden balance instrument 50 centimeters long, 4 centimeters high and 3 centimeters wide. He bends his other foot from his knee and holds it with his hand on the same side. While the patient is in balance with one foot in this way, the time begins and tries to stay in balance for 1 minute. The time is stopped when the balance is disturbed (leaving it while holding the foot, falling from the board to the ground, touching the ground with any part of its body, etc.). When the patient goes up to the balance device and restores his balance, the time continues from where he left off. The test continues for a minute. When the time is completed, each patient's attempt to balance (after falling) is counted, and this number is recorded as the patient's score at the end of the test when one minute has been completed.
One Leg Stand Test | Change from baseline to 8 weeks, follow up at two months
  It is a test in which the patient's right and left extremity is measured in balance time and evaluates the static balance. If the patient can stand on one foot for 180 seconds, the test is considered complete. In our study, one foot standing test will be performed in accordance with the criteria specified in the literature. Patients are asked to stand as much as possible on one foot with their eyes open and in a standing position, and the time they are stopped is measured in seconds, measured by a stopwatch. An experiment is made before registration and then the test is repeated 3 times. No oral stimuli are given during the test. The stopwatch is stopped when the patient's foot in the air touches the ground or when the patient loses his standing position (47). Static balance assessment of the cases will be evaluated by standing on one leg test.
Bioelectrical Impedance Analysis | Change from baseline to 8 weeks, follow up at two months
  The method is based on the difference between the lean tissue mass and the electrical permeability of the oil. In the method, weak electrical current impedance is measured. Hand-to-hand, hand-to-foot, foot-to-foot measurements can be made with different BIA analysis tools. Many other data are obtained, such as the amount of body fat, lean body mass, body water, and the distribution of fat in various parts of the body. It is a practical, easy to use and recommended method. The muscle, fat and water ratio of the cases will be evaluated with the InBody Bioelectric Impedance Device.
PostureScreen Mobile | Change from baseline to 8 weeks, follow up at two months
  There are different systems that use digital photographs and software analysis in posture evaluation. PostureScreen Mobile (posture analysis / body composition / motion evaluation software) is a valid and reliable application developed to evaluate posture with the help of a camera system on devices with iOS and Android systems. Posture evaluation is done through the program using the PostureScreen Mobile application. On the front and side photographs of the individual, the specific points determined in the software are marked using the touch screen, and according to these points, the values of the postural disorder and the degree of the disorder are calculated and reported for each patient in "centimeters" by software. Posture evaluation of the cases will be done with PostureScreen Mobile.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)